CLINICAL TRIAL: NCT03012126
Title: Childhood Obesity Research Demonstration Project 2.0 (CORD 2.0)
Brief Title: Clinical & Community Approaches to Weight Management
Acronym: CORD 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Department of Health (Other Government); Y-USA (Unknown); Yale University (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Chief, Division of General Academic Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 937121
Record Dates: First submitted 2016-12-12; First posted 2017-01-06 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Children were randomized to either: 1) federally qualified health center-based Healthy Weight Clinic, or 2) YMCA community-based Healthy Weight and Your Child Program.
  A comparison sample of children receiving care in eight demographically similar FQHCs serve as a comparison group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinically Based: Healthy Weight Clinic (Experimental): All families referred to the Healthy Weight Clinic intervention arm will be scheduled for a 30-45 minute orientation clinic visit to orient the child and family to the program. During this visit, the family will meet with the community health worker who will provide a schedule of clinic visits and dietitian contacts. The community health worker will assess the child's social and environmental context to allow treatment tailoring. For the first 6 months, each family will be asked to attend two clinic visits per month and complete weekly 20-30 minute contacts with the dietitian via telephone. The program aims to deliver approximately 30 contact hours in the 6-month period. This will be followed by monthly visits to the Healthy Weight Clinic and monthly calls with their dietitian.
  Interventions: Behavioral: Healthy Weight Clinic
- Community Based: Healthy Weight & Your Child (Experimental): All families referred to the Healthy Weight and Your Child intervention arm will be scheduled for a 60-minute family information session to orient the child and family to the program. During this visit, the family will receive information about the program and logistics such as program schedule and format and attendance. The program is delivered over 12 months, which includes 16 weekly sessions, followed by 4 sessions delivered every other week and concluding with 5 monthly sessions. Most sessions are 2 hours in length and include a group of about 8-15 children and their caregivers. The first hour is delivered in a classroom setting and the second hour in an additional area conducive for physical activity.
  Interventions: Behavioral: Healthy Weight and Your Child

INTERVENTIONS:
Behavioral: Healthy Weight Clinic
  Arms: Clinically Based: Healthy Weight Clinic
Behavioral: Healthy Weight and Your Child
  Arms: Community Based: Healthy Weight & Your Child

SUMMARY:
This project seeks to build on innovative strategies to optimize the care of low-income children with a BMI ≥ 85th percentile. To accomplish this goal, investigators will implement a new clinical-community intervention, theoretically grounded in the Integrated Clinical and Community Systems of Care Model, to address obesity through optimized screening and management known to be effective, e-Referrals, Healthy Weight Clinics, and the YMCA's Healthy Weight and Your Child weight management program (originally known as MEND). The study will examine outcomes for children that matter most to a broad group of stakeholders including parents, clinicians, and public health practitioners as well as inform the care of >7 million children with obesity covered by the Children's Health Insurance Program or Medicaid.

DETAILED DESCRIPTION:
This is a 2-arm RCT. Enrolled patients are randomized to a pediatric weight management intervention (PWMI): 1)a Healthy Weight Clinic based at a federally-qualified health center (FQHC), or 2) a modified Healthy Weight and Your Child intervention delivered in YMCAs. A comparison sample of children receiving care in eight demographically similar FQHCs serve as a comparison group.

ELIGIBILITY:
Inclusion Criteria:

* child is age 6.0 through 12.9 years at referral
* child's BMI meets or exceeds the 85th percentile for age and sex
* parent can read and respond to interviews and questionnaires in English and Spanish

Exclusion Criteria:

* children who do not have at least one parent who is able to follow study procedures for 1 year
* families who plan to leave their primary care health center within the study time frame
* families for whom the primary care clinician thinks the intervention is inappropriate, e.g., emotional or cognitive difficulties
* children who were taking medications that substantially interfere with growth
* children who have a sibling enrolled in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 407 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in Child BMI at 12 months | 0-12 months
Change in Child BMI percent of the 95th percentile at 12 months | 0-12 months

SECONDARY OUTCOMES:
Change in Screen Time at 12 months | 0-12 months
  Average hours per day of screen time as reported by parent
Change in Sleep Duration at 12 months | 0-12 months
  Average hours per day of sleep as reported by parent
Change in Physical Activity at 12 months | 0-12 months
  Average number of days (0-7) child is physically active for at least 60 minutes as reported by parent
Change in Diet at 12 months | 0-12 months
  Average daily intake of sugar-sweetened beverages and weekly intake of fast food as reported by parent

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Taveras, MD, MPH, Principal Investigator — MassGeneral Hospital for Children

IPD SHARING:
Plan to Share IPD: Yes
Individual-level data may be shared upon request, under the conditions that an analysis plan is prepared and approved by the PI/Co-Is, IRB approval has been obtained, and all necessary data sharing agreements have been executed.
Supporting Information: Study Protocol
Time Frame: Data can be requested by emailing the PI or Project Manager.
Access Criteria: 1. An analysis plan is prepared and approved by the PI/Co-Is
  2. IRB approval has been obtained, and
  3. all necessary data sharing agreements have been executed.

REFERENCES:
- [Background] Fiechtner L, Perkins M, Biggs V, Langhans N, Sharifi M, O'Connor G, Price S, Locascio J, Kuhlthau K, Kwass JA, Nelson C, Land T, Longjohn M, Lawson V, Hohman K, Taveras EM. Rationale and design of the Clinic and Community Approaches to Healthy Weight Randomized Trial. Contemp Clin Trials. 2018 Apr;67:16-22. doi: 10.1016/j.cct.2018.01.002. Epub 2018 Jan 10. PMID 29330083
- [Derived] Fay C, Castro I, Sierra Velez D, Ruggiero CF, O'Connor G, Perkins M, Luo M, Sharifi M, Neri Mini F, Taveras EM, Kuhlthau K, Fiechtner L. Keys to Achieving Clinically Important Weight Loss: Perceptions of Responders and Nonresponders in the Clinic and Community Approaches to Healthy Weight Trial. Child Obes. 2023 Dec;19(8):507-514. doi: 10.1089/chi.2022.0112. Epub 2022 Oct 28. PMID 36315223
- [Derived] Harshman SG, Castro I, Perkins M, Luo M, Barrett Mueller K, Cena H, Portale S, Raspini B, Taveras E, Fiechtner L. Pediatric weight management interventions improve prevalence of overeating behaviors. Int J Obes (Lond). 2022 Mar;46(3):630-636. doi: 10.1038/s41366-021-00989-x. Epub 2021 Dec 3. PMID 34862470
- [Derived] Sierra Velez D, Simione M, Castro I, Perkins M, Luo M, Taveras EM, Fiechtner L. Effects of a Pediatric Weight Management Intervention on Parental Stress. Child Obes. 2022 Apr;18(3):160-167. doi: 10.1089/chi.2021.0146. Epub 2021 Oct 7. PMID 34619054
- [Derived] Fiechtner L, Perkins M, Biggs V, Langhans N, Sharifi M, Price S, Luo M, Locascio JJ, Hohman KH, Hodge H, Gortmaker S, Torres S, Taveras EM. Comparative Effectiveness of Clinical and Community-Based Approaches to Healthy Weight. Pediatrics. 2021 Oct;148(4):e2021050405. doi: 10.1542/peds.2021-050405. Epub 2021 Sep 1. PMID 34470816
- [Derived] Atkins M, Castro I, Sharifi M, Perkins M, O'Connor G, Sandel M, Taveras EM, Fiechtner L. Unmet Social Needs and Adherence to Pediatric Weight Management Interventions: Massachusetts, 2017-2019. Am J Public Health. 2020 Jul;110(S2):S251-S257. doi: 10.2105/AJPH.2020.305772. PMID 32663093